CLINICAL TRIAL: NCT06316882
Title: ROGCAS - Retrospective Observational Gastric Cancer Study
Brief Title: Gastric Cancer Endoscopic Screening in an Intermediate-risk Country - ROGCAS, a Dual-centre Pilot Program
Acronym: ROGCAS
Status: Completed | Type: Observational
Sponsor: Unidade Local De Saúde Do Norte Alentejano (Other)
Collaborators: NOVA Medical School (Other); Universidade Nova de Lisboa (Other)
Responsible Party: Principal Investigator, Beatriz Mourato, Principal Investigator, Universidade Nova de Lisboa
Other Study IDs: ROGCAS
Record Dates: First submitted 2023-11-21; First posted 2024-03-19 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer; Gastric (Stomach) Cancer; Atrophic Gastritis; Intestinal Metaplasia of Gastric Mucosa; HELICOBACTER PYLORI INFECTIONS; High Grade Intraepithelial Neoplasia
Keywords: Gastric Cancer; Endoscopic screening; intermediated risk countries
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- screening endoscopy: We perform upper endoscopy, when the patient authorizes it, at the same time of their screening colonoscopy
  Interventions: Diagnostic Test: Screening endoscopy

INTERVENTIONS:
Diagnostic Test: Screening endoscopy — We perform upper endoscopy, when the patient authorizes it, during their screening colonoscopy
  Other Names: upper endoscopy

SUMMARY:
Endoscopic screening of gastric cancer combined with screening colonoscopy

DETAILED DESCRIPTION:
This is an observational retrospective research entitled "Gastric cancer endoscopic screening in an intermediate-risk country - ROGCAS, a dual-centre pilot program" (STROBE protocol. This study will analyze the results of an initiative of the ULSAALE Endoscopy Units, which, with the approval of the Board of Directors and Ethics Committee, started an opportunistic screening pilot program for oesophagogastric cancer in February 2023, inviting users from the national colorectal screening program to undergo EGD at the same time as screening colonoscopy. Based on the assumptions of the theoretical models of cost-effectiveness studies, we will analyze the efficacy of endoscopic screening for GC by determining the HP infection rate, the pre-malignant lesion detection rate, the GC detection rate, the early GC detection rate, the stage at diagnosis, the adherence rate and the cost of this pilot program. This study will be carried out in the Endoscopy Units of Hospital Doutor José Maria Grande and Hospital de Santa Luzia de Elvas, with the approval of the Board of Directors and the Ethics Committee of ULSAALE, and data will be collected by consulting the Sclinico records of patients who agree to participate in the study and who have undergone EGD and screening colonoscopy at the same time in these hospitals. In terms of potential benefits, this study could help to elucidate the appropriateness of introducing endoscopic GC screening at the same time as colorectal cancer screening in order to detect pre-malignant and malignant lesions at an earlier stage, thus improving the management and prognosis of this pathology.

On the other hand, users can undergo two endoscopic screenings simultaneously with the same sedation, saving time and resources and reducing the number of referrals to health centers. In terms of risks, there are those associated with endoscopic procedure and those associated with the screening process. As for complications, although rare, bleeding, perforation and infection have been described, but ULSAALE has expert teams of gastroenterologists and surgeons to deal with these complications. There are also risks associated with the sedation process, related to local and systemic pharmacological reactions and the possible need for ventilatory support, which is why an anaesthesiologist and/or an advanced life support team is always present. The risks of the screening program itself are related to false positive results and overdiagnosis. False positives, in addition to the potential psychological damage to the patient, lead to unnecessary diagnostic investigations and consumption of resources. Overdiagnosis, on the other hand, could place a burden on health services, both in terms of surveillance of premalignant lesions and in terms of providing timely treatment to patients diagnosed with GC. However, since this is a pathology with a high incidence and mortality rate in Portugal, the benefits of early diagnosis and improved prognosis seem to outweigh the inherent risks of the endoscopic screening program. Participation in this study is also voluntary and all participants will be asked to give informed consent after receiving adequate information and personal reflection.

ELIGIBILITY:
Inclusion Criteria:

* people who agree to undergo endoscopic screening for gastric cancer;
* people who undergo screening colonoscopy

Exclusion Criteria:

* Exams without biopsies

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people proposed to undergo colonoscopy to screen for colorectal cancer after a positive fecal occult blood test, through the national colorectal cancer screening program and who agreed to undergo endoscopy to screen for esophagogastric lesions
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
number of gastric adenocarcinoma | 1 month
  number of gastric adenocarcinomas detected in patients undergoing opportunistic endoscopic screening, confirmed by histological examination of biopsies obtained during the screening endoscopic examination

SECONDARY OUTCOMES:
number of pre-malignant lesions | 1 month
  number of cases of intestinal metaplasia or atrophic gastritis detected in the histological examination of biopsies obtained during endoscopic screening
Costs of screening endoscopy | 1 year
  costs in euros of each endoscopic examination in addition to the base cost of the scheduled colonoscopy screening
Socio-demographic characteristics of population in screening program | 1 month
  Determine the correlation between the socio-demographic characteristics of patients and the detection of gastric cancer by opportunistic screening

CONTACTS AND LOCATIONS:
Locations (1):
- ULSNA, Portalegre, Portalegre District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Endoscopic images; endoscopy reports; histopathology reports
Supporting Information: Study Protocol, CSR
Time Frame: end of study
Access Criteria: investigators of other clinical trials and systematic reviews

REFERENCES:
- [Background] Januszewicz W, Turkot MH, Malfertheiner P, Regula J. A Global Perspective on Gastric Cancer Screening: Which Concepts Are Feasible, and When? Cancers (Basel). 2023 Jan 21;15(3):664. doi: 10.3390/cancers15030664. PMID 36765621
- [Background] Areia M, Spaander MC, Kuipers EJ, Dinis-Ribeiro M. Endoscopic screening for gastric cancer: A cost-utility analysis for countries with an intermediate gastric cancer risk. United European Gastroenterol J. 2018 Mar;6(2):192-202. doi: 10.1177/2050640617722902. Epub 2017 Jul 18. PMID 29511549
- [Background] Faria L, Silva JC, Rodriguez-Carrasco M, Pimentel-Nunes P, Dinis-Ribeiro M, Libanio D. Gastric cancer screening: a systematic review and meta-analysis. Scand J Gastroenterol. 2022 Oct;57(10):1178-1188. doi: 10.1080/00365521.2022.2068966. Epub 2022 May 9. PMID 35531944
- [Background] Kim H, Hwang Y, Sung H, Jang J, Ahn C, Kim SG, Yoo KY, Park SK. Effectiveness of Gastric Cancer Screening on Gastric Cancer Incidence and Mortality in a Community-Based Prospective Cohort. Cancer Res Treat. 2018 Apr;50(2):582-589. doi: 10.4143/crt.2017.048. Epub 2017 Jun 9. PMID 28602053
- [Background] Rawla P, Barsouk A. Epidemiology of gastric cancer: global trends, risk factors and prevention. Prz Gastroenterol. 2019;14(1):26-38. doi: 10.5114/pg.2018.80001. Epub 2018 Nov 28. PMID 30944675
- [Background] Lopez MJ, Carbajal J, Alfaro AL, Saravia LG, Zanabria D, Araujo JM, Quispe L, Zevallos A, Buleje JL, Cho CE, Sarmiento M, Pinto JA, Fajardo W. Characteristics of gastric cancer around the world. Crit Rev Oncol Hematol. 2023 Jan;181:103841. doi: 10.1016/j.critrevonc.2022.103841. Epub 2022 Oct 11. PMID 36240980
- [Background] Kim GH, Liang PS, Bang SJ, Hwang JH. Screening and surveillance for gastric cancer in the United States: Is it needed? Gastrointest Endosc. 2016 Jul;84(1):18-28. doi: 10.1016/j.gie.2016.02.028. Epub 2016 Mar 3. PMID 26940296
- [Background] Lansdorp-Vogelaar I, Meester RGS, Laszkowska M, Escudero FA, Ward ZJ, Yeh JM. Cost-effectiveness of prevention and early detection of gastric cancer in Western countries. Best Pract Res Clin Gastroenterol. 2021 Mar-Apr;50-51:101735. doi: 10.1016/j.bpg.2021.101735. Epub 2021 Feb 22. PMID 33975689
- [Background] Almeida N, Romaozinho JM, Donato MM, Luxo C, Cardoso O, Cipriano MA, Marinho C, Fernandes A, Calhau C, Sofia C. Helicobacter pylori antimicrobial resistance rates in the central region of Portugal. Clin Microbiol Infect. 2014 Nov;20(11):1127-33. doi: 10.1111/1469-0691.12701. Epub 2014 Jul 12. PMID 24890952
- [Background] He J, Hu W, Ouyang Q, Zhang S, He L, Chen W, Li X, Hu C. Helicobacter pylori infection induces stem cell-like properties in Correa cascade of gastric cancer. Cancer Lett. 2022 Aug 28;542:215764. doi: 10.1016/j.canlet.2022.215764. Epub 2022 May 31. PMID 35654291
- [Background] Leja M, You W, Camargo MC, Saito H. Implementation of gastric cancer screening - the global experience. Best Pract Res Clin Gastroenterol. 2014 Dec;28(6):1093-106. doi: 10.1016/j.bpg.2014.09.005. Epub 2014 Sep 28. PMID 25439074
- [Background] Burra P, Bretthauer M, Buti Ferret M, Dugic A, Fracasso P, Leja M, Matysiak Budnik T, Michl P, Ricciardiello L, Seufferlein T, van Leerdam M, Botos A. Digestive cancer screening across Europe. United European Gastroenterol J. 2022 May;10(4):435-437. doi: 10.1002/ueg2.12230. Epub 2022 Apr 26. No abstract available. PMID 35474447
- [Background] Saftoiu A, Hassan C, Areia M, Bhutani MS, Bisschops R, Bories E, Cazacu IM, Dekker E, Deprez PH, Pereira SP, Senore C, Capocaccia R, Antonelli G, van Hooft J, Messmann H, Siersema PD, Dinis-Ribeiro M, Ponchon T. Role of gastrointestinal endoscopy in the screening of digestive tract cancers in Europe: European Society of Gastrointestinal Endoscopy (ESGE) Position Statement. Endoscopy. 2020 Apr;52(4):293-304. doi: 10.1055/a-1104-5245. Epub 2020 Feb 12. PMID 32052404
- [Background] Areia M, Carvalho R, Cadime AT, Rocha Goncalves F, Dinis-Ribeiro M. Screening for gastric cancer and surveillance of premalignant lesions: a systematic review of cost-effectiveness studies. Helicobacter. 2013 Oct;18(5):325-37. doi: 10.1111/hel.12050. Epub 2013 Apr 9. PMID 23566268
- [Background] Ishii N, Shiratori Y, Ishikane M, Omata F. Population effectiveness of endoscopy screening for mortality reduction in gastric cancer. DEN Open. 2023 Sep 19;4(1):e296. doi: 10.1002/deo2.296. eCollection 2024 Apr. PMID 37731836
- [Derived] Mourato MB, Pratas N, Branco Pereira A, Costa Pinto F, Dinis R, Fronteira I, Areia M. Gastric Cancer Endoscopic Screening in an Intermediate-Risk Country-A Dual-Center Pilot Program. Helicobacter. 2025 Jul-Aug;30(4):e70061. doi: 10.1111/hel.70061. PMID 40762368
- See also: Global Cancer Observatory — https://gco.iarc.fr/today/online-analysis-map?v=2020&mode=population&mode_population=continents&population=900&populations=900&key=asr&sex=0&cancer=7&type=0&statistic=5&prevalence=0&population_group=0&ages_group%5B%5D=0&ages_group%5B%5D=17&nb_items=10&group_cancer=1&include_nmsc=0&include_nmsc_other=0&projection=natural-earth&color_palette=default&map_scale=quantile&map_nb_colors=5&continent=0&show_ranking=0&rotate=%255B10%252C0%255D
- See also: National Cancer Institute — https://portal.gdc.cancer.gov